CLINICAL TRIAL: NCT03489291
Title: Phase IIb, Open-label, Single-dose, Single-arm, Multi-center Trial to Confirm the Factor IX Activity Level of the Serotype 5 Adeno-associated Viral Vector Containing the Padua Variant of a Codon-optimized Human Factor IX Gene (AAV5-hFIXco-Padua, AMT-061) Administered to Adult Subjects With Severe or Moderately Severe Hemophilia B
Brief Title: Dose Confirmation Trial of AAV5-hFIXco-Padua
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSL222_2001 (CT-AMT-061-01)
Record Dates: First submitted 2018-03-19; First posted 2018-04-05 (Actual); Results first posted 2022-06-16 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Hemophilia B
Keywords: Hemophilia,; Gene Therapy; Bleeding; Factor IX; FIX; viral vector; Padua
MeSH Terms: conditions — Hemophilia B; Hemophilia A; Hemorrhage

STUDY DESIGN:
Intervention Model Description: open-label, single-dose, single-arm, multi-center trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single infusion of AMT-061 (Experimental): Subjects will receive a single infusion of AAV5-hFIXco-Padua (AMT- 061) at baseline. After IMP administration (post IMP), subjects will be monitored for tolerance to the IMP and detection of potential immediate AEs at the clinical trial site for 24 hours (overnight stay).
  Interventions: Genetic: AAV5-hFIXco-Padua (AMT-061)

INTERVENTIONS:
Genetic: AAV5-hFIXco-Padua (AMT-061) — Single intravenous infusion of AAV5-hFIXco-Padua (AMT-061)

SUMMARY:
This is an open-label, single-dose, single-arm, multi-center trial, with a screening, a treatment + post-treatment follow-up phase, and a long-term follow-up phase.

The IMP AMT-061 is a recombinant adeno-associated viral vector of serotype 5 (AAV5) containing the Padua variant of a codon-optimized human FIX complementary deoxyribonucleic acid (cDNA) under the control of a liver-specific promoter. The IMP is identified as AAV5-hFIXco-Padua (AMT- 061). The pharmaceutical form of AMT-061 is a solution for intravenous infusion.

The administered dose of AMT-061 will be 2 x 10^13 gc/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age ≥18 years
3. Subjects with congenital hemophilia B classified as severe or moderately severe
4. >20 previous exposure days of treatment with FIX protein

Exclusion Criteria:

1. History of FIX inhibitors
2. Positive FIX inhibitor test at screening
3. Select screening laboratory values > 2 times upper normal limit:
4. Positive human immunodeficiency virus (HIV) at screening, not controlled with anti-viral therapy
5. Active infection with Hepatitis B or C virus at screening
6. History of Hepatitis B or C exposure, currently controlled by antiviral therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Hemophilia B is an X-linked, recessive condition, since it occurs almost exclusively in males. Females typically are asymptomatic carriers. Therefore eligibility is restricted to male participants.
Enrollment: 3 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2023-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Pipe, MD, Principal Investigator — University of Michigan
Locations (4):
- United States (4):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of California, Davis, Sacramento, California
  - University of California, San Diego, San Diego, California
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] von Drygalski A, Gomez E, Giermasz A, Castaman G, Key NS, Lattimore SU, Leebeek FWG, Miesbach WA, Recht M, Monahan PE, Le Quellec S, Pipe SW. Completion of phase 2b trial of etranacogene dezaparvovec gene therapy in patients with hemophilia B over 5 years. Blood Adv. 2025 Jul 22;9(14):3543-3552. doi: 10.1182/bloodadvances.2024015291. PMID 40188458
- [Derived] O'Connell N, van der Valk P, Le Quellec S, Gomez E, Monahan PE, Crary SE, Coppens M, Lemons R, Castaman G, Klamroth R, Symington E, Quon DV, Kampmann P. Invasive procedures and surgery following etranacogene dezaparvovec gene therapy in people with hemophilia B. J Thromb Haemost. 2025 Jan;23(1):73-84. doi: 10.1016/j.jtha.2024.08.027. Epub 2024 Sep 26. PMID 39341368
- [Derived] von Drygalski A, Gomez E, Giermasz A, Castaman G, Key NS, Lattimore SU, Leebeek FWG, Miesbach WA, Recht M, Gut R, Dolmetsch R, Monahan PE, Le Quellec S, Pipe SW. Stable and durable factor IX levels in patients with hemophilia B over 3 years after etranacogene dezaparvovec gene therapy. Blood Adv. 2023 Oct 10;7(19):5671-5679. doi: 10.1182/bloodadvances.2022008886. PMID 36490302
- [Derived] Von Drygalski A, Giermasz A, Castaman G, Key NS, Lattimore S, Leebeek FWG, Miesbach W, Recht M, Long A, Gut R, Sawyer EK, Pipe SW. Etranacogene dezaparvovec (AMT-061 phase 2b): normal/near normal FIX activity and bleed cessation in hemophilia B. Blood Adv. 2019 Nov 12;3(21):3241-3247. doi: 10.1182/bloodadvances.2019000811. PMID 31698454

RESULTS

PARTICIPANT FLOW:
Groups:
- AMT-061 (CSL222): Adeno-associated viral vector serotype 5 (AAV5)-hFIXco-Padua (AMT-061 [CSL222]): Single intravenous infusion of AMT-061 (CSL222).
Period: Overall Study
Arm/Group | AMT-061 (CSL222)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- AMT-061 (CSL222): AAV5-hFIXco-Padua (AMT-061 [CSL222]): Single intravenous infusion of AMT-061 (CSL222).
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Factor IX Activity Levels
Description: To confirm that a single dose of 2x10^13 gc/kg AMT-061 (CSL222) resulted in factor IX activity levels of ≥5% at 6 weeks after dosing measured by the one-stage (activated partial thromboplastin [aPTT]-based) assay.
Time Frame: 6 weeks post-dose
Population: All subjects treated.
Measure: Mean (Standard Deviation); unit: Factor IX activity (%)
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Factor IX activity (%) | 30.6 (6.97)

2. Secondary Outcome: Annualized Exogenous Factor IX Usage
Description: Annualized use was calculated as the normalized amount of therapy administered per baseline weight, extrapolated where necessary from any time period less or greater than 1 year. Therapy administered included the total dosage of FIX given as prophylaxis and on-demand. Use for invasive procedures was not included.
Time Frame: 52 weeks post-dose
Population: All subjects treated.
Measure: Mean (Standard Deviation); unit: International units (IU)/kg/year
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
International units (IU)/kg/year | 7.1 (6.4)

3. Secondary Outcome: Annualized Bleeding Rate (ABR)
Description: ABR was calculated as the ratio of the number of bleeds to the number of days in the time interval multiplied by 365.25.
Time Frame: 5 years post-dose
Population: All subjects treated.
Measure: Number; unit: bleeds/year/subject
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
bleeds/year/subject
  All bleeds (Spontaneous + Traumatic + Joint) | 0.14
  Spontaneous bleeds | 0.07
  Traumatic bleeds | 0.07
  Joint bleeds | 0.00

4. Secondary Outcome: Factor IX Activity Levels
Description: Measured by the one-stage (aPTT-based) assay.
Time Frame: 52 weeks post-dose
Population: All subjects treated.
Measure: Mean (Standard Deviation); unit: Factor IX activity (%)
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Factor IX activity (%) | 40.8 (9.45)

5. Secondary Outcome: Number of Participants Remaining Free of Continuous Prophylaxis
Description: Participants with no usage of continuous factor IX prophylaxis after AMT-061 (CSL222) treatment were considered free from continuous factor IX prophylaxis use.
Time Frame: 1 year post-dose
Population: All subjects treated.
Measure: Count of Participants; unit: Participants
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Participants | 3

6. Secondary Outcome: Annualized Exogenous Factor IX Usage Post-Continuous Prophylaxis
Description: The post-continuous-prophylaxis period began on the day after the end of continuous (routine) prophylaxis.Therapy administered included the total dosage of FIX given as prophylaxis and on-demand. Use for invasive procedures was not included.
Time Frame: Up to 5 years post-dose
Population: All subjects treated.
Measure: Mean (Standard Deviation); unit: IU/year
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
IU/year | 342.1 (592.5)

7. Secondary Outcome: Number of Participants With Treatment Emergent (TE): Adverse Events (AE), Mild, Moderate, and Severe AEs, AEs Related and Unrelated to the Study Treatment, and Serious AEs
Time Frame: Up to 5 years post-dose
Population: All subjects treated.
Measure: Count of Participants; unit: Participants
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Participants
  Participant with TEAEs | 3
  Participant with mild TEAEs | 3
  Participant with moderate TEAEs | 2
  Participant with severe TEAEs | 2
  Participants with TEAEs related to study treatment | 1
  Participants with TEAEs unrelated to study treatment | 3
  Participants with serious TEAEs | 1

8. Secondary Outcome: Number of Participants With Clinically Meaningful Findings in Hematology and Serum Chemistry Parameters
Description: Clinically meaningful findings were defined as values which were outside the standard normal reference ranges for hematology and serum chemistry parameters.
Time Frame: Up to 5 years post-dose
Population: All subjects treated.
Measure: Count of Participants; unit: Participants
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Participants | 0

9. Secondary Outcome: Number of Participants With Newly Occurring or Worsening Potentially Clinically Significant Changes in Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) Levels
Description: Post-baseline newly occurring or worsening potentially clinically significant ALT and AST levels were defined as values greater than twice the baseline value.
Time Frame: From baseline and up to 5 years post-dose
Population: All subjects treated.
Measure: Count of Participants; unit: Participants
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Participants
  AST | 1
  ALT | 1

10. Secondary Outcome: Number of Participants Receiving Corticosteroids for AST and ALT Elevations
Time Frame: Up to 5 years post-dose
Population: All subjects treated.
Measure: Count of Participants; unit: Participants
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Participants | 0

11. Secondary Outcome: Number of Participants Positive With AAV5 and Factor IX Neutralising Antibodies in Serum
Time Frame: Baseline and at 5 years post-dose
Population: All subjects treated.
Measure: Count of Participants; unit: Participants
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Participants
  At Baseline for AAV5 | 3
  At 5 years post dose for AAV5 | 3
  At Baseline for FIX | 0
  At 5 years post dose for FIX | 0

12. Secondary Outcome: Number of Participants With AAV5 Capsid-specific T Cell Response
Time Frame: Up to Week 52
Population: All subjects treated.
Measure: Count of Participants; unit: Participants
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Participants | 1

13. Secondary Outcome: Number of Participants With Inflammatory Marker Levels Outside Normal Ranges
Description: Inflammatory markers included interleukin (IL)-1β, IL-2, IL-6, interferon gamma (IFNγ), and monocyte chemotactic protein-1 (MCP-1). Only those biomarkers for which the data were higher than the normal range at the specified timepoints have been presented.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16, 18, 20, 22, 24, 26, 31, 36, 40, 44, 48 and 52
Population: All subjects treated.
Measure: Count of Participants; unit: Participants
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Participants
  Baseline: MCP-1 | 1
  Week 1: MCP-1 | 1
  Week 8: MCP-1 | 1
  Week 40: IL-6 | 1

14. Secondary Outcome: Time to First Negative Results for Vector Deoxyribonucleic Acid (DNA) From Semen and Blood
Description: Time in weeks until the first negative result confirmed by negative result in 3 consecutive timepoints. A participant was considered to no longer be shedding vector DNA if they had a negative laboratory result for 3 or more consecutive timepoints.
Time Frame: Up to 5 years post-dose
Population: All subjects treated. Here, the "Number Analyzed (n)" included participants who were evaluable at specific parameters.
Measure: Median (Full Range); unit: Weeks
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Weeks
  Semen: number analyzed (Participants) | 2
  Semen | 26.21 [26.1 to 26.3]
  Blood | 78.29 [31.1 to 168.9]

15. Secondary Outcome: Number of Participants With Abnormal Values in Alpha-fetoprotein (AFP) Levels
Description: Participants who were outside the normal limit range were to be reported.
Time Frame: Up to 5 years post-dose
Population: All subjects treated.
Measure: Count of Participants; unit: Participants
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Participants | 0

16. Secondary Outcome: Number of Participants With Abnormal Results in Abdominal Ultrasound
Description: Ultrasounds were evaluated by qualified personnel and abnormalities were assessed by the Investigator.
Time Frame: At Months 36, 42, 48, 54, and 60 post-dose
Population: All subjects treated. Here, the "Number Analyzed (n)" included participants who were evaluable at specific timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Participants
  Month 36 | 3
  Month 42: number analyzed (Participants) | 2
  Month 42 | 2
  Month 48 | 3
  Month 54 | 2
  Month 60 | 3

17. Post Hoc Outcome: Factor IX Activity Levels
Description: To confirm that a single dose of 2x10^13 gc/kg AMT-061 (CSL222) resulted in factor IX activity levels of ≥5% at 5 years after dosing measured by the one-stage (activated partial thromboplastin [aPTT]-based) assay.
Time Frame: 5 years post dose
Population: All subjects treated.
Measure: Mean (Standard Deviation); unit: Factor IX activity (%)
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Factor IX activity (%) | 45.67 (6.18)

18. Post Hoc Outcome: Number of Participants Remaining Free of Continuous Prophylaxis
Description: as for outcome 5
Time Frame: 5 years post dose
Population: All subjects treated.
Measure: Count of Participants; unit: Participants
Arm/Group | AMT-061 (CSL222)
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: 5 years post-dose
Arm/Group | AMT-061 (CSL222)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMT-061 (CSL222) (N=3)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMT-061 (CSL222) (N=3)
Bronchitis (Infections and infestations) | 1 (1)
COVID 19 (Infections and infestations) | 1 (1)
Coccidioidomycosis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (3)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (5)
Dizziness (Nervous system disorders) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 1 (2)
Paraesthesia (Nervous system disorders) | 1 (2)
Sciatica (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (2)
Dental caries (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (3)
Tongue disorder (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (3)
Chronic fatigue syndrome (General disorders) | 1 (1)
Pain (General disorders) | 1 (6)
Alanine aminotransferase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
C reactive protein increased (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Amblyopia (Eye disorders) | 1 (1)
Cataract nuclear (Eye disorders) | 1 (1)
Pinguecula (Eye disorders) | 1 (1)
Pseudophakia (Eye disorders) | 1 (1)
Refraction disorder (Eye disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (2)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Peripheral coldness (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT03489291/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT03489291/SAP_001.pdf